CLINICAL TRIAL: NCT05475379
Title: A Randomized Control, Double Blinded, Non-inferiority Trial to Evaluate the Immunogenicity and Safety of Typhoid Vi Conjugate Vaccine 'Typhocon' in Bangladeshi Healthy Population
Brief Title: Non-inferiority Trial of Locally Manufactured Typhoid Conjugate Vaccine 'Typhocon' in Bangladesh
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PR-22013
Record Dates: First submitted 2022-06-11; First posted 2022-07-26 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2022-07

CONDITIONS: Typhoid
Keywords: Conjugate vaccine; Immunogenicity; Safety; Typhoid fever
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a randomized double-blind study. Study investigators along with study staff involved in safety evaluation and laboratory analysis will be blinded regarding the assigned treatment of the participant. The vaccine administration team will be un-blinded to the treatment assignment list. The vaccine administrator team members will not be involved in the evaluation of vaccine safety and laboratory analysis. The DSMB will be responsible for un-blinding the randomization number codes in the event of severe putative vaccine reactions. Otherwise, the codes will not be revealed until the end of the trial and until the computerized dataset has been frozen. If the intervention assignment is un-blinded, all study collaborators will be notified immediately. If deemed necessary, the DSMBs will recommend unblinding to the IRB and contact the study statistician responsible for providing information on the vaccine received by the individual in question.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test vaccine group (Experimental): 300 participants will receive Typhoid Vi polysaccharide-diphtheria toxoid conjugate vaccine (Vi-DT)
  Trade name: Typhocon®, Incepta Vaccine Ltd.
  Interventions: Biological: Typhoid Vi polysaccharide-diphtheria toxoid conjugate vaccine (Vi-DT)
- Reference vaccine group (Active Comparator): 300 participants will receive Vi polysaccharide-tetanus toxoid conjugate vaccine (Vi-TCV)
  Trade name: Typbar-TCV®, Bharat-Biotech International Limited.
  Interventions: Biological: Typhoid Vi polysaccharide-diphtheria toxoid conjugate vaccine (Vi-DT)

INTERVENTIONS:
Biological: Typhoid Vi polysaccharide-diphtheria toxoid conjugate vaccine (Vi-DT) — Typhoid Vi-polysaccharide-diphtheria toxoid conjugate vaccine (Vi-DT) "Typhocon" will be manufactured by Incepta Vaccine Limited
  Other Names: Vi polysaccharide-tetanus toxoid conjugate vaccine (Vi-TCV)

SUMMARY:
This is a double blinded, randomized-controlled, non-inferiority trial of a typhoid conjugate vaccine, Typhocon (Vi- polysaccharide conjugated to diphtheria toxoid, Vi-DT), manufactured by a local company, Incepta Vaccine Limited. The vaccine will be tested among individuals from 6 months to 60 years of age residing in Mirpur area of Dhaka city. The Typbar-TCV (Vi-polysaccharide conjugated to tetanus toxoid, Vi-TT), manufactured by Bharat Biotech International Limited will be used as a reference vaccine in this study.

In Phase I the Typhocon vaccine will be tested in 30 adults. Safety and immunogenicity data of the vaccine for 30 adults will be submitted to the Data Safety Monitoring Board (DSMB), IRB and Directorate General of Drug Administration (DGDA). Upon receiving approval letter, the investigators will initiate the Phase II study including 600 individuals. The Phase II study will be conducted in age de-escalation manner (6-23 months, 2-5 years, 6-17 years and 18-60 years). Equal number of participants of all age groups will be enrolled for vaccination. Blood specimens will also be collected for carrying out the clinical chemistry (complete blood count with differential for white blood count, hemoglobin, absolute neutrophil count, platelet count, serum alanine transaminase, serum creatinine) on day -7 to day -2 for screening of participants before vaccination and on day 28, postvaccination. Based on blood reports of clinical chemistry, 600 participants will be randomized in a 1:1 ratio to allocate Typhocon or Typbar-TCV vaccine. Memory aid will be used to collect solicited adverse events following vaccination (AEFI) data up to day 7. Data on unsolicited AEFI and serious adverse events (SAEs) will be collected up to 28 days after vaccination. All study update including adverse events and serious adverse events will be reported to the DSMB. Blood specimen will be obtained on day 0 before vaccination, and day 28 for carrying out Enzyme-linked Immunosorbent Assay (ELISA) to determine anti-Vi-IgG antibody.

DETAILED DESCRIPTION:
A double blinded, randomized-controlled, non-inferiority trial of a typhoid conjugate vaccine, Typhocon (Vi- polysaccharide conjugated to diphtheria toxoid, Vi-DT), manufactured by a local company, Incepta Vaccine Limited will be conducted. The vaccine will be tested among individuals from 6 months to 60 years of age residing in Mirpur area of Dhaka city. The Typbar-TCV (Vi-polysaccharide conjugated to tetanus toxoid, Vi-TT), manufactured by Bharat Biotech International Limited will be used as a reference vaccine in this study.

Hypothesis:

Locally produced typhoid conjugate vaccine 'Typhocon' is non-inferior in terms of safety and immunogenicity among healthy Bangladeshi population as compared to 'Typbar-TCV'.

Objectives:

1. To evaluate and compare the safety of locally produced 'Typhocon' with 'Typbar- TCV'.
2. To evaluate and compare the immunogenicity of 'Typhocon' with 'Typbar-TCV' in healthy population in Bangladesh.

   Number of participants for enrollment:

   Age group Test vaccine Reference vaccine 18-60 Years 75 75 6-17 Years 75 75 2-5 Years 75 75 6-23 Months 75 75 Total 300 300

   Study activities:

   Screening and eligibility assessment:

   Study field staff will visit different households in Mirpur area and brief apparently healthy and eligible participants about the study. They will invite them to Mirpur field clinic to be included as participants in the study. If agreed, written consent will be obtained from the participants at the field clinic. Blood specimens will be collected for carrying out clinical chemistry (complete blood count with differential for white blood count, hemoglobin, absolute neutrophil count, platelet count, serum alanine transaminase, serum creatinine). Participants with abnormalities in screening hematological and biochemical tests will be excluded for vaccination. After screening, the eligible participant will be enrolled for vaccination after matching with inclusion and exclusion criteria. A study ID will be provided to each participant once informed written consent has been obtained.

   Informed consent:

   The participants/parent/guardian must personally sign and date the latest approved version of the Informed Consent form before any trial specific procedures are performed. Assent will also be sought from children 11-17 years of age or older, to participate in the trial. Consent will be documented by signature or thumbprint on consent forms. Participants will read the informed consent or that will be read out to the ones who are not literate, and they will be encouraged to ask questions regarding the study. Informed consent will be obtained from participants who agree to take vaccine and give blood at two time points during the study period. Signature (or thumbprint, if illiterate) of each of the participants will be obtained before their enrollment in the study and prior to any study-related activity. A witness and the study personnel who obtains the consent must sign and date in the informed consent form. The participant will be provided with a copy of the signed consent form for their retention.

   If new information is obtained which is not covered in the proposal on the study product but becomes available later on and is relevant to the participants' willingness to continue in the study, the investigator will inform that in a timely manner to the IRB and use a revised written informed consent form. The proposal will be revised and resubmitted to RRC and ERC for the amendment which will then be used for obtaining permission. The clinical trial will be monitored by the sponsor.

   Randomisation:

   The randomization for this study will be generated using the statistical software. Each participant will be assigned with unique participant ID. The study agents (Typhocon or Typbar-TCV) will be labelled by Incepta Vaccine Limited as per the randomization list and the list will be provided by them. Randomization sheet will contain sequential treatment numbers unique to each participant.

   Blinding and Code Breaking Procedures:

   This is a randomized double-blind study. Study investigators along with study staff involved in safety evaluation and laboratory analysis will be blinded regarding the assigned treatment of the participant. The vaccine administration team will be un-blinded to the treatment assignment list. The vaccine administrator team members will not be involved in the evaluation of vaccine safety and laboratory analysis. The DSMB will be responsible for un-blinding the randomization number codes in the event of severe putative vaccine reactions. Otherwise, the codes will not be revealed until the end of the trial and until the computerized dataset has been frozen. If the intervention assignment is un-blinded, all study collaborators will be notified immediately. If deemed necessary, the DSMBs will recommend unblinding to the IRB and contact the study statistician responsible for providing information on the vaccine received by the individual in question.

   Vaccination of participants:

   Potential participants will attend the vaccination site. Upon arrival, inclusion/exclusion criteria will be assessed, and written informed consent/assent will be formally obtained with the participants/parent/ guardian of the participant. The participant will then be vaccinated, and a blood sample will be taken for immunological assay before vaccination. All details will be recorded in the CRF. Based on the randomization, the appropriate vaccine will be administered by a trained member of the study team. The site of vaccination (right or left arm or thigh) will be recorded.

   Investigational Product:

   Test vaccine: Typhocon (Incepta Vaccine Limited) Reference vaccine: Typbar-TCV (Bharat Biotech International Limited)

   Dosage and administration:

   For children and adults, the same dose (0.5 ml) of vaccine in prefilled syringe will be administered via intramuscular route on day 0 will be given.

   Visit 1: Day -7 to -2 Screening:

   The following procedures will be followed after obtaining the informed consent from the participants to determine the eligibility for participating in the study. At the screening visit(s), the designated study staff will provide a detailed description of the study objectives to the participant and also describe study participation requirements, potential health risks and benefits associated with study participation.
   1. Written informed consent will be obtained and any remaining questions that the participant may have will be solicited/discussed.
   2. A participant ID number will be assigned once the study specific consent form has been signed.
   3. Demographic information will be obtained.
   4. Vital signs (Blood pressure, pulse rate, respiratory rate and temperature) will be recorded.
   5. Medical history will be obtained and a thorough physical examination will be performed by a physician. In addition, medical history will be taken thoroughly by study physician from the woman of childbearing age to completely exclude the probability of pregnancy during screening and prior to vaccination. Women who are married and living with a partner must agree to use a reliable contraceptive method to prevent pregnancy until final follow-up following vaccination. However abstinence is also acceptable.
   6. Inclusion/exclusion criteria are reviewed to determine qualification for enrollment, including medications used in the past 30 days.
   7. Females with child bearing potential, a urine dipstick pregnancy test will be performed and verified as negative prior to phlebotomy.
   8. Blood samples (3-10ml) will be collected for Complete Blood Count (CBC) with differential for white blood count (WBC), hemoglobin (Hg) , Absolute Neutrophil Count (ANC), platelet count, Serum Alanine Transaminase (ALT), Serum Creatinine for screening of participants to enroll in the study. Plasma/serum will be separated from blood to determine anti-Vi-IgG antibody response for vaccinees.

   Visit-2: Day: 0 Enrollment and vaccination:
   1. Clinical evaluation and eligibility criteria will be reviewed by study physician to determine qualification for enrollment, including medications. Vital signs (Blood pressure, pulse rate, respiratory rate and temperature) will be recorded.
   2. Females with child bearing potential, a urine dipstick pregnancy test will be performed and verified as negative prior to vaccination.
   3. The study agent (Typhocon or Typbar-TCV) will be given to the participant intramuscularly according to the randomization.
   4. The participants will be observed for 30 minutes for solicited reactogenicity symptoms.
   5. Vital signs (Blood pressure, pulse rate, respiratory rate and temperature) will be checked at least 30 minutes post-dose.
   6. Each participant will be provided with a memory aid to record solicited symptoms on a daily basis through Day 7. Participants will be trained to record temperature and any symptoms on the memory aid.
   7. Study staff will instruct the participant regarding continued assessment of his/her health and need to contact study staff (a) for follow-up of specific AEs, (b) if systemic symptoms worsen or do not resolve, and (c) if other AEs occur.
   8. Participants will be instructed to bring the memory aid to the next scheduled clinic visit.
   9. The next visit for Day 7 will be instructed. The vaccine will be administered by a trained study nurse. During vaccination, a team of trained doctors, nurses and medical technologists will be available at the vaccination sites to deal with all emergency situation including anaphylaxis. To deal with anaphylaxis first-line and second-line equipment will be available whenever a vaccine is administered at the vaccination sites. These will be physically separated into two separate boxes. Both boxes will be clearly labeled and kept together.

   The essential first-line equipment is to be used by any staff member trained in anaphylaxis and basic life support. It includes the following:
   * Adrenaline: at least 2 x 1ml vials of 1:1000 (1mg/mL)
   * Filter needles
   * 1ml syringes
   * Needles for IM injection: 25mm (23G) is appropriate
   * Cotton wool/gauze
   * Pocket masks (facemasks) for BLS
   * Paediatric and adult sizes
   * Copy of treatment algorithm
   * Copy of adrenaline dosage table
   * List of emergency contact numbers

   The essential second-line equipment is only to be used by trained medical personnel, such as doctors. It includes the following:
   * Self-inflating resuscitation bag (as part of a bag-valve-mask system)
   * 500ml for infants up to around 2 years
   * 1600ml - 2000ml for older children
   * Masks compatible with bag
   * Include 3 to 4 sizes, suitable sizes for infants to adults
   * Chlorphenamine: solution for injection, minimum of 10mg
   * For example 1 x 1ml vial of 10mg/ml solution
   * Hydrocortisone: solution for injection, minimum of 200For example 2 x 1ml vials of 100mg/ml solution
   * Salbutamol: dry powder inhaler, 100microgram per dose
   * Spacer for use with inhaler
   * Filter needles
   * 1ml syringes
   * 5ml syringes
   * Needles for IM injection: 25mm is appropriate
   * Cotton wool/gauze
   * Copy of advanced (second-line) treatment algorithm
   * Copy of drug dosage tables
   * List of emergency contact numbers

   Visit-3: Day: 7 (+3) Memory aid collection:

   The investigators will collect parent/guardian-reported information on adverse events following immunization (AEFIs). The investigators will encourage the parents/guardians to visit field clinic if any adverse event happens other than the schedule visit.

   Visit-4: Day: 28 (+7) Follow-up:
   1. Participants will visit field clinic for clinical evaluation.
   2. Blood samples (3-10ml) will be collected for Complete Blood Count (CBC) with differential for white blood count (WBC), hemoglobin (Hg) , Absolute Neutrophil Count (ANC), platelet count, Serum Alanine Transaminase (ALT), Serum Creatinine for clinical chemistry. Plasma/serum will be separated from blood to determine anti-Vi-IgG antibody response for vaccinees.

   Visit-5: Day: 90 (±7) Follow-up:

   The participant will come to Mirpur Field clinic and physical examination with vital sign (blood pressure, respiratory rate, pulse rate and temperature) will be performed.

   Laboratory assay:

   Blood samples will be transported to the laboratory to processed and stored by trained study staff, in accordance with standard operating procedures (SOP). The plasma/serum will be stored and used to measure the induced immune response in the vaccinees. The primary laboratory technique performed will be anti-Vi antibody ELISA performed on the extracted plasma sample, using a commercially available assay (VaccZyme, The Binding Site). This assay will be performed according to the manufacturer's instructions.

   Investigational Medicinal Product (IMP):

   IMP description Test vaccine

   Typhoid Vi polysaccharide-diphtheria toxoid conjugate vaccine (Vi-DT). Trade name: Typhocon®, Incepta Vaccine Ltd.

   Each 0.5ml vaccine dose contains:
   * Purified Typhoid Conjugate Bulk: 25 µg
   * Sodium Chloride: 8.7 mg
   * Disodium Hydrogen Phosphate Heptahydrate: 2.34 mg
   * Sodium Dihydrogen Phosphate Monohydrate: 0.23 mg

   Reference vaccine

   Vi polysaccharide-tetanus toxoid conjugate vaccine (Vi-TCV). Trade name: Typbar-TCV®, Bharat-Biotech International Limited.

   Each 0.5ml vaccine dose contains:
   * Purified Vi-Capsular Polysaccharide of S. Typhi Ty2 conjugated to Tetanus Toxoid 25µg
   * Sodium chloride 4.5 mg
   * Water for Injection q.s. to 0.5ml

   The vaccine is packaged as a pre-filled syringe and the Strength is 25 µg/0.5 ml. It will be administered as an intramuscular injection in the antero-lateral thigh for younger children, or the upper arm for older children, according to local protocols.

   Supply:

   Both test (Typhocon) and reference (Typbar-TCV) vaccines will be provided by Incepta vaccine limited.

   Storage:

   The vaccines will be stored at 2o to 8o C (35 o to 46 o F) in a temperature monitored cold room at the icddr,b, when not in use for the daily activities. The vaccines will be stored in temperature monitored refrigerators or cool boxes, when in use for the day's activities. Each vial will be labelled with a "vaccine vial monitor"; a temperature-sensitive dot that provides an indication of the cumulative heat to which the vial has been exposed. It warns the end user when exposure to heat is likely to have degraded the vaccine beyond an acceptable level and should not be used.

   Accountability of the trial treatment:

   The vaccines will be shipped to a central storage facility in the icddr,b. They will then be transported and distributed to the vaccine site whilst maintaining the cold-chain (aiming for temperature between 2-8oC).

   The number of doses of study vaccines that are received, used and wasted will be documented daily during the trial and checked weekly.

   Procedures for recording adverse events

   From vaccination through day 7:

   All adverse events related to vaccination, as judged by a medically qualified investigator, occurring during the first 7 days post vaccination that are observed by the study team/investigator or reported by the participants' parent/guardian, will be recorded on the CRF. The information will be collected both passively and actively. Parents of participants not in this subset will be encouraged to go to the 'Adverse Event Monitoring Cell' at the Mirpur Field Clinic which will have a medical doctor on-call 24 hours a day for adverse event monitoring throughout the whole vaccination period + 7 days.

   The following information will be recorded: description, date of onset and end date, severity, assessment of relatedness to trial medication, and action taken. Follow-up information should be provided as necessary.

   The severity of events will be assessed on the following scale: 1 = mild, 2 = moderate, 3 = severe.

   All Serious Adverse Events (SAEs) observed by the Investigator, members of the study team or reported by the parent/guardian will be recorded on the CRF.

   The following information will be recorded: description, date of onset and end date, severity, assessment of relatedness to trial medication, other suspect drug or device and action taken. Follow-up information should be provided as necessary.

   Throughout the study period:

   Serious Adverse Events (SAEs), as judged by a medically qualified investigator, observed by the Investigator, members of the study team or reported by the parent/guardian, will be recorded on the CRF.

   The following information will be recorded: description, date of onset and end date, severity, assessment of relatedness to trial medication, and action taken. Follow-up information should be provided as necessary.

   All mortality occurring during the duration of the trial will be recorded in the CRF, and investigated by medically qualified trial staff.

   All SAEs recorded in the CRFs, for the duration of the study, from first vaccination until trial completion, will be followed by a medically qualified investigator either until resolution, or until the event is considered stable.

   Reporting procedures for serious adverse events:

   For this study, forms will be used for reporting all SAEs occurring during this study.

   All SAEs occurring within the first 30 days, post vaccine administration, and then only SARs occurring until the end of the trial, will be reported to the Data Safety Monitoring Board (DSMB), Directorate General of Drug Administration (DGDA), the PI and the other study Investigators within 24 hours of the Site Study Team becoming aware of the event. A more detailed report form will be completed during medical follow-up, and sent within the shortest period possible of the initial report, to all parties mentioned above. Additional and further requested information (follow-up or corrections to the original case) will be detailed in subsequent safety report forms. All SAEs must be reported to the trial sponsor within 7 days.

   Summary reports will be submitted to the icddr,b IRB, and DGDA at the end of the study. SAEs will also be reported to the sponsor.

   Sample size calculation and outcome:

   Primary outcome of this study is the seroconversion rate (4-fold rise of anti-Vi plasma/serum immunoglobulin G (IgG) enzyme-linked immunosorbent assay titers over baseline). For the sample size calculation, the investigators are assuming 85% seroconversion rates for both reference (Typbar-TCV) and test (Typhocon) vaccines at day 28 after vaccination. The difference of seroconversion rates as large as 10% in favor of Typhocon vaccine would still allow to be non-inferior at 10% margin (delta = 0.10). To confirm non-inferiority with 90% study power and a one-sided confidence level of 97.5%, the investigators will need at least 270 study participants for each arm (total 540). Anticipating 10% attrition rate, the investigators will enroll total 600 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed written consent from participants or if minor from their parent/legal guardian
2. Healthy participants aged 6 months to 60 years
3. Family does not have any plan to move from the study area during study period.

Exclusion Criteria:

1. History of hypersensitivity reaction to any component of the study vaccines.
2. History of typhoid vaccination within the last three years.
3. Fever of any origin or infections of more than 3 days within the past month.
4. Subjects with febrile illness (temperature >37.9 C) at the time of enrollment.
5. History of any vaccination within the past 30 days.
6. Clinically significant systemic disorder such as cardiovascular, respiratory, neurologic, gastrointestinal, hepatic, renal, endocrine, hematological or immunological disorder.
7. Participants with abnormalities in screening hematological and biochemical tests will be excluded for vaccination
8. Subjects with confirmed or suspected immunosuppressive or immunodeficiency disorder; or subjects on any immunosuppressive or immunostimulant therapy.
9. Known case of thrombocytopenia or any coagulation disorder, or subjects on anticoagulation therapy.
10. Subjects administered blood, blood containing products or immunoglobulins within the last 3 months or planned administration during the study.
11. Urine dipstick pregnancy test verified as positive
12. Pregnant* and lactating women & female subjects not using acceptable contraceptive measures (double barrier methods, oral or injectable hormonal contraceptives or surgical sterilization).

    * Urine pregnancy test (UPT) will be performed in all married females prior to vaccination

Ages: 6 Months to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 630 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants developing adverse events and serious adverse events | 28 days
  Proportion of participants developing adverse events following immunization (AEFI) and serious adverse events (SAE). To estimate the proportion of safety data, the investigators will use memory aid, and AEFI and SAE forms to collect the data.

SECONDARY OUTCOMES:
Immune response induced in vaccinees | 6 months
  To measure the immune response induced in vaccinees, blood specimens will be collected. Plasma/serum will be separated from blood specimens and anti Vi-IgG antibody responses will be measured using the commercially available kit.

CONTACTS AND LOCATIONS:
Overall Officials: Farhana Khanam, MPhil, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crump JA, Luby SP, Mintz ED. The global burden of typhoid fever. Bull World Health Organ. 2004 May;82(5):346-53. PMID 15298225
- [Background] Antillon M, Warren JL, Crawford FW, Weinberger DM, Kurum E, Pak GD, Marks F, Pitzer VE. The burden of typhoid fever in low- and middle-income countries: A meta-regression approach. PLoS Negl Trop Dis. 2017 Feb 27;11(2):e0005376. doi: 10.1371/journal.pntd.0005376. eCollection 2017 Feb. PMID 28241011
- [Background] Meiring JE, Shakya M, Khanam F, Voysey M, Phillips MT, Tonks S, Thindwa D, Darton TC, Dongol S, Karkey A, Zaman K, Baker S, Dolecek C, Dunstan SJ, Dougan G, Holt KE, Heyderman RS, Qadri F, Pitzer VE, Basnyat B, Gordon MA, Clemens J, Pollard AJ; STRATAA Study Group. Burden of enteric fever at three urban sites in Africa and Asia: a multicentre population-based study. Lancet Glob Health. 2021 Dec;9(12):e1688-e1696. doi: 10.1016/S2214-109X(21)00370-3. PMID 34798028
- [Background] World Health Organization. Typhoid vaccines: WHO position paper, March 2018 - Recommendations. Vaccine. 2019 Jan 7;37(2):214-216. doi: 10.1016/j.vaccine.2018.04.022. Epub 2018 Apr 13. PMID 29661581
- [Background] Qamar FN, Yousafzai MT, Khaliq A, Karim S, Memon H, Junejo A, Baig I, Rahman N, Bhurgry S, Afroz H, Sami U. Adverse events following immunization with typhoid conjugate vaccine in an outbreak setting in Hyderabad, Pakistan. Vaccine. 2020 Apr 23;38(19):3518-3523. doi: 10.1016/j.vaccine.2020.03.028. Epub 2020 Mar 20. PMID 32201138
- [Background] Mohan VK, Varanasi V, Singh A, Pasetti MF, Levine MM, Venkatesan R, Ella KM. Safety and immunogenicity of a Vi polysaccharide-tetanus toxoid conjugate vaccine (Typbar-TCV) in healthy infants, children, and adults in typhoid endemic areas: a multicenter, 2-cohort, open-label, double-blind, randomized controlled phase 3 study. Clin Infect Dis. 2015 Aug 1;61(3):393-402. doi: 10.1093/cid/civ295. Epub 2015 Apr 13. PMID 25870324
- [Background] Qadri F, Khanam F, Liu X, Theiss-Nyland K, Biswas PK, Bhuiyan AI, Ahmmed F, Colin-Jones R, Smith N, Tonks S, Voysey M, Mujadidi YF, Mazur O, Rajib NH, Hossen MI, Ahmed SU, Khan A, Rahman N, Babu G, Greenland M, Kelly S, Ireen M, Islam K, O'Reilly P, Scherrer KS, Pitzer VE, Neuzil KM, Zaman K, Pollard AJ, Clemens JD. Protection by vaccination of children against typhoid fever with a Vi-tetanus toxoid conjugate vaccine in urban Bangladesh: a cluster-randomised trial. Lancet. 2021 Aug 21;398(10301):675-684. doi: 10.1016/S0140-6736(21)01124-7. Epub 2021 Aug 9. PMID 34384540
- [Background] Theiss-Nyland K, Shakya M, Colin-Jones R, Voysey M, Smith N, Karkey A, Dongol S, Pant D, Farooq YG, Neuzil KM, Shrestha S, Basnyat B, Pollard AJ. Assessing the Impact of a Vi-polysaccharide Conjugate Vaccine in Preventing Typhoid Infections Among Nepalese Children: A Protocol for a Phase III, Randomized Control Trial. Clin Infect Dis. 2019 Mar 7;68(Suppl 2):S67-S73. doi: 10.1093/cid/ciy1106. PMID 30845329
- [Background] Patel PD, Patel P, Liang Y, Meiring JE, Misiri T, Mwakiseghile F, Tracy JK, Masesa C, Msuku H, Banda D, Mbewe M, Henrion M, Adetunji F, Simiyu K, Rotrosen E, Birkhold M, Nampota N, Nyirenda OM, Kotloff K, Gmeiner M, Dube Q, Kawalazira G, Laurens MB, Heyderman RS, Gordon MA, Neuzil KM; TyVAC Malawi Team. Safety and Efficacy of a Typhoid Conjugate Vaccine in Malawian Children. N Engl J Med. 2021 Sep 16;385(12):1104-1115. doi: 10.1056/NEJMoa2035916. PMID 34525285
- [Background] Mond JJ, Lees A, Snapper CM. T cell-independent antigens type 2. Annu Rev Immunol. 1995;13:655-92. doi: 10.1146/annurev.iy.13.040195.003255. PMID 7612238
- [Background] Weintraub A. Immunology of bacterial polysaccharide antigens. Carbohydr Res. 2003 Nov 14;338(23):2539-47. doi: 10.1016/j.carres.2003.07.008. PMID 14670715
- [Background] Acharya IL, Lowe CU, Thapa R, Gurubacharya VL, Shrestha MB, Cadoz M, Schulz D, Armand J, Bryla DA, Trollfors B, et al. Prevention of typhoid fever in Nepal with the Vi capsular polysaccharide of Salmonella typhi. A preliminary report. N Engl J Med. 1987 Oct 29;317(18):1101-4. doi: 10.1056/NEJM198710293171801. PMID 3657877
- [Background] Klugman KP, Gilbertson IT, Koornhof HJ, Robbins JB, Schneerson R, Schulz D, Cadoz M, Armand J. Protective activity of Vi capsular polysaccharide vaccine against typhoid fever. Lancet. 1987 Nov 21;2(8569):1165-9. doi: 10.1016/s0140-6736(87)91316-x. PMID 2890805
- [Background] Yang HH, Wu CG, Xie GZ, Gu QW, Wang BR, Wang LY, Wang HF, Ding ZS, Yang Y, Tan WS, Wang WY, Wang XC, Qin M, Wang JH, Tang HA, Jiang XM, Li YH, Wang ML, Zhang SL, Li GL. Efficacy trial of Vi polysaccharide vaccine against typhoid fever in south-western China. Bull World Health Organ. 2001;79(7):625-31. PMID 11477965
- [Background] Froeschle JE, Decker MD. Duration of Vi antibodies in participants vaccinated with Typhim Vi (Typhoid Vi polysaccharide vaccine) in an area not endemic for typhoid fever. Vaccine. 2010 Feb 10;28(6):1451-3. doi: 10.1016/j.vaccine.2009.11.051. Epub 2009 Dec 8. PMID 20003920
- [Background] Michel R, Garnotel E, Spiegel A, Morillon M, Saliou P, Boutin JP. Outbreak of typhoid fever in vaccinated members of the French Armed Forces in the Ivory Coast. Eur J Epidemiol. 2005;20(7):635-42. doi: 10.1007/s10654-005-7454-6. PMID 16119438
- [Background] Pasetti MF, Simon JK, Sztein MB, Levine MM. Immunology of gut mucosal vaccines. Immunol Rev. 2011 Jan;239(1):125-48. doi: 10.1111/j.1600-065X.2010.00970.x. PMID 21198669
- [Background] Cryz SJ Jr, Vanprapar N, Thisyakorn U, Olanratmanee T, Losonsky G, Levine MM, Chearskul S. Safety and immunogenicity of Salmonella typhi Ty21a vaccine in young Thai children. Infect Immun. 1993 Mar;61(3):1149-51. doi: 10.1128/iai.61.3.1149-1151.1993. PMID 8432597
- [Background] Simanjuntak CH, Paleologo FP, Punjabi NH, Darmowigoto R, Soeprawoto, Totosudirjo H, Haryanto P, Suprijanto E, Witham ND, Hoffman SL. Oral immunisation against typhoid fever in Indonesia with Ty21a vaccine. Lancet. 1991 Oct 26;338(8774):1055-9. doi: 10.1016/0140-6736(91)91910-m. PMID 1681365
- [Background] Levine MM, Ferreccio C, Black RE, Germanier R. Large-scale field trial of Ty21a live oral typhoid vaccine in enteric-coated capsule formulation. Lancet. 1987 May 9;1(8541):1049-52. doi: 10.1016/s0140-6736(87)90480-6. PMID 2883393
- [Background] Olanratmanee T, Levine M, Losonsky G, Thisyakorn V, Cryz SJ Jr. Safety and immunogenicity of Salmonella typhi Ty21a liquid formulation vaccine in 4- to 6-year-old Thai children. J Infect Dis. 1992 Aug;166(2):451-2. doi: 10.1093/infdis/166.2.451. No abstract available. PMID 1634818